CLINICAL TRIAL: NCT03369314
Title: Observational, Real-life Study of the Use of octaplasLG®.
Brief Title: Observational Study of the Use of octaplasLG®.
Status: Completed | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: TMA POOL
Record Dates: First submitted 2017-11-30; First posted 2017-12-12 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Receiving octaplasLG®: The data will be collected in all patients who have received at least one infusion of octaplasLG®
  Interventions: Drug: octaplasLG®

INTERVENTIONS:
Drug: octaplasLG® — Data will be collected in all patients who have received at least one infusion of octaplasLG®

SUMMARY:
This observational study enrolls patients who have received at least one infusion of octaplasLG®. OctaplasLG® will be administered standard of care and observation occurs during the treatment and 24 hours after the end of treatment. Characteristics of the use of octaplasLG®, tolerance criteria, and efficacy criteria will be collected.

DETAILED DESCRIPTION:
Prospective, non-interventional, multicentre study meeting a post-marketing need. The data will be collected in all patients who have received at least one infusion of octaplasLG®.

The duration of follow-up is limited to the duration of treatment with octaplasLG® plus 24 h of monitoring after cessation of treatment.

Characteristics of the use of octaplasLG® (indication for the transfusion, degree of urgency, characteristics of plasma infusions, patient characteristics, number of iso-group and/or compatible units administered, tolerance criteria (adverse effects), and efficacy criteria (for patients with confirmed diagnosis of TTP--time to normalization of platelet count) will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is treated with octaplasLG® (receiving at least 1 unit of 200 ml octaplasLG®)
2. In accordance with Reference Methodology MR-003, the patient of legal age must be individually informed through an information sheet, and must not oppose participating in this non-interventional study (with no collection of consent). If the patient is unable to receive the information and express any opposition, family members or the trusted person receive the information and must not oppose the collection of data*. For minor patients, one of the holders of parental authority receive the information and must not oppose the collection of data.

   * However, the patient in question will be informed if his/her condition later allows.

Exclusion Criteria:

1) Patient's refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Analyses will be carried out on all patients included, i.e. who have received at least one unit of octaplasLG®. This population will be stratified based on the different product indications.
  For the population defined as that of patients with TTP, only those patients for whom the investigator has indicated a confirmed diagnosis of idiopathic TTP will be included in the efficacy analysis (see secondary objective).
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Indication for the transfusion of octaplasLG® | From start of treatment to 24 hours following treatment with octaplasLG®
  Indication for the transfusion of octaplasLG®
Degree of urgency - Ordering department of octaplasLG® | From start of treatment to 24 hours following treatment with octaplasLG®
  Degree of urgency - Ordering department of octaplasLG®
Characteristics of the plasma infusions performed (transfusion or PE, administration rate, volume, date) | From start of treatment to 24 hours following treatment with octaplasLG®
  Characteristics of the plasma infusions performed (transfusion or PE, administration rate, volume, date)
Patient characteristics (socio-demographic criteria, blood group, dominant pathology, co-morbidities including allergies, prior treatments) | From start of treatment to 24 hours following treatment with octaplasLG®
  Patient characteristics (socio-demographic criteria, blood group, dominant pathology, co-morbidities including allergies, prior treatments)
Number of iso-group and/or compatible units administered for octaplasLG® | From start of treatment to 24 hours following treatment with octaplasLG®
  Number of iso-group and/or compatible units administered for octaplasLG®

SECONDARY OUTCOMES:
Tolerance of octaplasLG®: Adverse effects (with notion of Severity and Imputability, time to onset/start of infusion) associated with the plasma | From start of treatment to 24 hours following treatment with octaplasLG®
  Tolerance of octaplasLG®: Adverse effects (with notion of Severity and Imputability, time to onset/start of infusion) associated with the plasma including allergic immunological type (e.g. TRALI) and other events (infections, related to the PE procedure (e.g. case of transfusion-associated circulatory overload [TACO], citrate reaction, etc.).
Efficacy criteria in the treatment of TTP including time to normalisation of platelet count (time between first PE procedure and a confirmed platelet count > 150 x 109/L on at least 2 consecutive days) | From start of treatment to 24 hours following treatment with octaplasLG®
  Efficacy criteria in the treatment of TTP including time to normalisation of platelet count (time between first PE procedure and a confirmed platelet count > 150 x 109/L on at least 2 consecutive days)

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CH Henri Duffaut, Avignon
  - Hôpital de La Cavale Blanche, Brest
  - Hôpital Louis Pradel, Bron
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Hospices Civils de Lyon Hôpital Edouard Herriot, Lyon
  - Hôpital de la Conception, Marseille
  - APHP Hopital Pitié salpêtrière, Paris
  - APHP Hopital Cochin, Paris
  - CHU Hôpitaux de Rouen, Rouen
  - CHRU Hôpital Nord, Saint-Etienne
  - Hôpital Foch, Suresnes
  - Clinique Pasteur, Toulouse
  - CHRU Bretonneau, Tours
  - CHU de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided